CLINICAL TRIAL: NCT06019949
Title: Neuromodulatory Rehabilitation for Respiratory Motor Function in Individuals With Chronic Spinal Cord Injury
Brief Title: Spinal Cord Stimulation for Respiratory Rehabilitation in Patients With Chronic Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Alexander V Ovechkin, MD, PhD, Assistant Professor, M.D., Ph.D., University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23.0570; 1R01HL168294 (NIH)
Record Dates: First submitted 2023-08-22; First posted 2023-08-31 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Spinal Cord Injuries; Respiration Disorders
Keywords: Spinal Cord Injury; Respiration; Rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries; Respiration Disorders; Respiratory Aspiration | interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: Thirty-six SCI participants will be randomly assigned to three groups (n=12 in each group): those who receive RT alone, scTS alone, or a combination of both (scTS+RT).
  After screening and recruitment, primary and secondary outcome measurements will be obtained in the Lab at the following time points: 1) Pre-intervention, after 30-days without any stimulation and/or intervention, 2) Post mapping, (participants with scTS), 3) Post Session #40 (after 8 weeks of intervention), 4) Post Session #80 (after 16 weeks of intervention), and 5) twice during 16-weeks Follow-up Period. In total, it is anticipated that 6 measurements will be obtained for each participant with scTS and 5 measurements for participants without scTS.
Who Masked: Outcomes Assessor
Masking Description: Unidentified data sets will be processed and evaluated by the research staff not directly involved in experimental procedures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Training (RT) group (Active Comparator): 80 scTS sessions will be administered using the Neostim/Biostim (Cosyma Inc., Denver CO) device applying up to five conductive electrodes placed on the skin at the midline over the thoracic levels as cathodes between T1 to T8, and up to four self-adhesive electrodes located symmetrically on the skin over the iliac crests and shoulders as anodes. During the intervention, optimally configured scTS will be delivered based on the measures assessed during mapping sessions. The scTS with 5 mA-sub-motor threshold intensity with optimal frequency and pulse width will be delivered using 5 min on and 5 min off stimulation periods during interventional bouts. Every research participant will be slowly acclimated to stimulation. Blood pressure, heart rate, and respiratory rate will be closely monitored throughout stimulation sessions in the Lab by using beat-to-beat blood pressure, and respiratory kinematics monitoring.
  Interventions: Device: Respiratory Training
- Spinal Cord Transcutaneous Stimulation (scTS) group (Active Comparator): Participants will undergo 80 RT sessions using standard threshold Positive Expiratory Pressure Device (PEP, Respironics Inc., Cedar Grove, NJ) and standard threshold Inspiratory Muscle Trainer (IMT, Respironics Inc., Cedar Grove, NJ) assembled together using a T-shaped connector with a flanged mouthpiece (Airlife 001504). Participants will be trained at the Frazier Rehab Institute and remotely to complete eighty 45-minute sessions during 16 weeks. The participants will be instructed to perform inspiratory and expiratory efforts against a pressure threshold load. The training will be initiated with a load equal to 20% of their individual Maximum Inspiratory Pressure (PImax) and Maximum Expiratory Pressure (PEmax) values with progressive increases as tolerated up to 60% of their baseline PImax and PEmax measures. The goal will be to reach the 60% load of PImax and PEmax during the last week of each month of the training.
  Interventions: Device: Transcutaneous spinal cord stimulator
- Spinal Cord Transcutaneous Stimulation and Respiratory Training (scTS+RT) group (Experimental): Participants will undergo 80 scTS combined with the RT while seated in their own wheelchairs with an approximately 45° head-up tilt. The scTS will be administered using the Neostim/Biostim (Cosyma Inc., Denver CO) and Standard threshold Positive Expiratory Pressure Device (PEP, Respironics Inc., Cedar Grove, NJ) and standard threshold Inspiratory Muscle Trainer (IMT, Respironics Inc., Cedar Grove, NJ) assembled together using a T-shaped connector with a flanged mouthpiece (Airlife 001504) will be used for the RT as described for the Arms 1 and 2.
  Interventions: Device: Transcutaneous spinal cord stimulator; Device: Respiratory Training

INTERVENTIONS:
Device: Transcutaneous spinal cord stimulator — Stimulation to the spinal cord will be administered using Neostim/Biostim (Cosyma Inc., Denver CO) device by applying up to five conductive electrodes placed on the skin at the midline over the thoracic levels as cathodes between T1 to T8, and up to four self-adhesive electrodes located symmetrically on the skin over the iliac crests and shoulders as anodes.
  Other Names: Non-invasive spinal cord stimulator
  Arms: Spinal Cord Transcutaneous Stimulation (scTS) group; Spinal Cord Transcutaneous Stimulation and Respiratory Training (scTS+RT) group
Device: Respiratory Training — Standard threshold Positive Expiratory Pressure Device (PEP, Respironics Inc., Cedar Grove, NJ) and standard threshold Inspiratory Muscle Trainer (IMT, Respironics Inc., Cedar Grove, NJ) assembled together using a T-shaped connector with a flanged mouthpiece (Airlife 001504) will be used for the respiratory training intervention.
  Other Names: Respiratory Muscle Training
  Arms: Spinal Cord Transcutaneous Stimulation and Respiratory Training (scTS+RT) group; Training (RT) group

SUMMARY:
Respiratory complications are among the leading causes of death in patients with chronic spinal cord injury (SCI). Our previous work showed that pulmonary function can be improved by using our original respiratory training method. However, the effectiveness of this intervention is limited due to the disruption of brain-spinal connections and consequently lowered spinal cord activity below the injury level. Our recent studies showed that electrical stimulation of the spinal cord below the level of injury leads to increased ventilation which indicates activation of the spinal cord structures related to respiration. These findings indicate that spinal cord stimulation can be a promising therapeutic additive to the treatment. The goal of this study is to justify the establishment of a new direction in rehabilitation for patients with SCI by using a non-invasive spinal cord stimulation in combination with respiratory training.

Our aims are: 1) to evaluate the effects of such stimulation applied to the injured spinal cord on pulmonary function and respiratory muscle activity, and 2) to evaluate the effectiveness and therapeutic mechanisms of the spinal cord stimulation combined with respiratory training. Thirty-six individuals with chronic SCI will be recruited and assigned to three groups to receive respiratory training or spinal cord stimulation alone or a combination of them. All participants will be tested before and after cycles of experimental procedures with/or without stimulation. Our hypotheses will be confirmed if the respiratory training combined with spinal cord stimulation results in the most enhanced positive effects.

DETAILED DESCRIPTION:
This is a respiratory rehabilitation-based clinical study consisting of physiologically and functionally relevant mapping of respiratory function that enhances our knowledge of neurophysiological modulation evoked by non-invasive spinal cord Transcutaneous Stimulation (scTS) and contributes to the development of the next generation of rehabilitative approaches. Following the screening process and recruiting, the research subjects will undergo the following procedures: Subjects (total n=36) will be randomly assigned to three groups and will undergo baseline assessments; evaluations before and after 80 sessions of specific intervention (Respiratory Training /RT/ alone, scTS alone, or RT in combination with scTS); and during 16 week-long follow up period.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old;
* stable medical condition;
* no painful musculoskeletal dysfunction, unhealed fracture, contracture, pressure sore or urinary tract infection that might interfere with respiratory training or stimulation;
* no clinically significant depression, psychiatric disorders or ongoing drug abuse;
* non-progressive SCI (no negative change in the neurological level and motor-completeness assessed during screening when compared to the neurological status assessed at 6-mo period after injury or at least 6 months prior to the screening), non-ventilator dependence, motor-complete SCI according to the American Spinal Injury Association Impairment Scale (AIS) grade "A" or "B" above T5 spinal level;
* sustained SCI at least 12 months prior to entering the study;
* compared to the normative values for healthy population, at least 15%-deficit in pulmonary function outcomes (FVC and FEV1) as detected by screening spirometry.

Exclusion Criteria:

Participants will be excluded from the study if there is a presence of

* major pulmonary or cardiovascular disease,
* ventilator dependence,
* endocrine disorders,
* malignancy,
* marked obesity,
* deep vein thrombosis,
* HIV/AIDS-related illness,
* secondary hypotension (anemia, hypervolemia, endocrine and neurological diseases),
* major esophageal/gastrointestinal problem or other major medical illness contraindicated for respiratory training or testing.

During screening, the potential participant will be asked whether she is pregnant or planning to become pregnant during the study period. Pregnant women are excluded from this study, as the risk to the fetus is unknown. No pregnancy test or birth control regimen will be required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-09-10 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2030-04-10 (Estimated)

PRIMARY OUTCOMES:
Maximum Expiratory Pressure (PEmax). | Within 2 weeks during screening period; within 4 weeks before an intervention period; within 2 weeks after intervention #40; within 2 weeks after intervention #80; within 2 weeks after 16-weeks and 32-weeks follow-up periods.
  Standard Spirometry measurement.
Maximum Inspiratory Pressure (PImax). | Within 2 weeks during screening period; within 4 weeks before an intervention period; within 2 weeks after intervention #40; within 2 weeks after intervention #80; within 2 weeks after 16-weeks and 32-weeks follow-up periods.
  Standard Spirometry measurement.
Surface electromyography (sEMG) Similarity Index (SI) | Within 4 weeks before an intervention period; within 2 weeks after intervention #40; within 2 weeks after intervention #80; within 2 weeks after 16-weeks and 32-weeks follow-up periods.
  Respiratory multi-muscle activation measures assessed using standard surface electromyography.

SECONDARY OUTCOMES:
Forced Vital Capacity (FVC). | Within 2 weeks during screening period; within 4 weeks before an intervention period; within 2 weeks after intervention #40; within 2 weeks after intervention #80; within 2 weeks after 16-weeks and 32-weeks follow-up periods.
  Standard Spirometry measurement.
Forced Expiratory Volume in 1 second (FEV1). | Within 2 weeks during screening period; within 4 weeks before an intervention period; within 2 weeks after intervention #40; within 2 weeks after intervention #80; within 2 weeks after 16-weeks and 32-weeks follow-up periods.
  Standard Spirometry measurement.
Baroreflex blood pressure sensitivity (BRS). | Within 4 weeks before an intervention period; within 2 weeks after intervention #40; within 2 weeks after intervention #80; within 2 weeks after 16-weeks and 32-weeks follow-up periods.
  Measure of the beat-to-beat blood pressure variability assessed during a Valsalva maneuver.
Baroreflex heart rate sensitivity (BRS). | Within 4 weeks before an intervention period; within 2 weeks after intervention #40; within 2 weeks after intervention #80; within 2 weeks after 16-weeks and 32-weeks follow-up periods.
  Measure of the beat-to-beat heart rate variability assessed during a Valsalva maneuver.
Baroreflex blood pressure effectiveness index (BEI). | Within 4 weeks before an intervention period; within 2 weeks after intervention #40; within 2 weeks after intervention #80; within 2 weeks after 16-weeks and 32-weeks follow-up periods.
  Measure of the beat-to-beat blood pressure variability assessed during a Valsalva maneuver.
Baroreflex heart rate effectiveness index (BEI). | Within 4 weeks before an intervention period; within 2 weeks after intervention #40; within 2 weeks after intervention #80; within 2 weeks after 16-weeks and 32-weeks follow-up periods.
  Measure of the beat-to-beat heart rate variability assessed during a Valsalva maneuver.
Spinal Cord Independence Measure (SCIM, Version III). | Within 4 weeks before an intervention period; within 2 weeks after intervention #40; within 2 weeks after intervention #80; within 2 weeks after 16-weeks and 32-weeks follow-up periods.
  Measures the level of self-care.

OTHER OUTCOMES:
The Craig Handicap Assessment & Reporting Technique (CHART) Questionnaire. | Within 4 weeks before an intervention period; within 2 weeks after intervention #40; within 2 weeks after intervention #80; within 2 weeks after 16-weeks and 32-weeks follow-up periods.
  Measures the level of handicap in a community setting.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Ovechkin, MD, PhD, Principal Investigator — University of Louisville
Locations (1):
- Frazier Rehabilitation and Neuroscience Institute, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No